CLINICAL TRIAL: NCT00724698
Title: Post-marketing Surveillance of the Safety, Tolerability and Efficacy of Desloratadine Tablet Among Filipino Patients
Brief Title: Evaluation of Desloratadine When Used in Patients With Either Allergic Rhinitis or Chronic Idiopathic Urticaria
Acronym: Aerius
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P04706
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2009-07-17 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis; Urticaria
MeSH Terms: conditions — Rhinitis; Urticaria | interventions — desloratadine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group: Patients diagnosed with Allergic Rhinitis or Chronic Idiopathic Urticaria
  Interventions: Drug: Desloratadine

INTERVENTIONS:
Drug: Desloratadine — Desloratadine 5 mg once daily
  Other Names: SCH 034117

SUMMARY:
Eligible patients will be prescribed Desloratadine 1 tablet of 5 mg once daily. Patients will be asked to follow-up for a final visit after 14 days (Day 15) where the safety, tolerability and clinical efficacy will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient men or women, age 12 years and above.
* Diagnosis of Allergic Rhinitis or Chronic Idiopathic Urticaria

Exclusion Criteria:

* Known hypersensitivity to Desloratadine.
* Pregnancy or lactation

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Filipino patients diagnosed to have Allergic Rhinitis or Chronic Idiopathic Urticaria
Sampling Method: Probability Sample
Enrollment: 3011 (Actual)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Desloratadine: Desloratadine 5 mg daily
Period: Overall Study
Arm/Group | Desloratadine
Started | 3011
Completed | 2921
Not Completed | 90
Not completed — Adverse Event | 9
Not completed — Failure of Therapy | 4
Not completed — Poor Compliance | 16
Not completed — Lost to Follow-up | 36
Not completed — No Info | 25

BASELINE CHARACTERISTICS:
Arm/Group | Desloratadine
Number analyzed (Participants) | 3011
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 239
  Between 18 and 65 years | 2542
  >=65 years | 230
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1788
  Male | 1223

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of adverse events reported
Time Frame: Final Visit (Day 15)
Measure: Number; unit: adverse events reported
Arm/Group | Desloratadine
Number analyzed (Participants) | 3011
adverse events reported
  Mild | 41
  Moderate | 15
  Severe | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agree only to use such information to conduct the study and will not be able to publish the results of any part of the study without previous writeen authorization from Schering-Plough.